CLINICAL TRIAL: NCT04956354
Title: The Use of Wireless Sensors in Neonatal Intensive Care (Wireless NICU)
Brief Title: The Use of Wireless Sensors in Neonatal Intensive Care
Status: Active, not recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Guilherme Sant'Anna, MD, Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: Wireless NICU
Record Dates: First submitted 2021-06-11; First posted 2021-07-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Preterm Birth; Apnea of Newborn
Keywords: Continuous monitoring; NICU; Wireless sensors
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Phase 1a: Once the setup of the study sensors is complete, clinical and physiological data will be continuously acquired for 8h during daytime, for 4 consecutive days. In addition, photographs of the skin at the site of placement of the sensors will be taken before sensors placement and after removal.
  Hourly axillary temperature measured by the bedside nurse (as part of routine care) will be manually recorded for each patient by the research team. A temperature and humidity recorder will also be placed around 15cm from the infants to continuously record air temperature and humidity.
  Interventions: Device: ANNE™ Monitoring System (2 sensors) - version B
- Phase 1b: Once the setup of the study sensors is complete, clinical and physiological data will be continuously acquired between 2h to 8h during daytime, for 2 to 4 consecutive days. In addition, photographs of the skin at the site of placement of the sensors will be taken before sensors placement and after removal.
  A temperature and humidity recorder will also be placed around 15cm from the infants to continuously record air temperature and humidity.
  Interventions: Device: ANNE™ Monitoring System (2 sensors) - version C
- Phase 2: Once the setup of the study sensors is complete, clinical and physiological data will be continuously acquired for a longer monitoring period - i.e., 96 consecutive hours. In consideration with device battery life, the devices will be replaced daily. In addition, photographs of the skin at the site of placement of the sensors will be taken at baseline, device replacement, and at 96h. The research team will also measure respirations using uncalibrated RIP belts at the level of the chest and abdomen (2 to 3 continuous hours each day). Two respiratory bands will be placed circumferentially around the infant's chest and around the abdomen to measure chest and abdominal wall movements, respectively.
  A temperature and humidity recorder will also be placed around 15cm from the infants to continuously record air temperature and humidity.
  Interventions: Device: ANNE™ Monitoring System (2 sensors) - version C

INTERVENTIONS:
Device: ANNE™ Monitoring System (2 sensors) - version B — ANNE™ is a wireless vital sign monitoring device that uses soft, flexible, skin-mountable biosensors (ANNE™ Chest and ANNE™ Limb) with Bluetooth® 5 enabled and encrypted data communication to an iPad application. Study sensors to be applied on patients are:
  Sensor 1 - A chest unit (ANNE™ Chest) with embedded battery, sensors, and a three-axis accelerometer that captures the following signals: electrocardiography (ECG), temperature, seismocardiography (SCG) and the chest wall movements.
  Sensor 2 - A limb unit (ANNE™ Limb) with embedded battery that captures the photoplethysmography (PPG) and SpO2 signals.
  Groups: Phase 1a
Device: ANNE™ Monitoring System (2 sensors) - version C — ANNE™ is a wireless vital sign monitoring device that uses soft, flexible, skin-mountable biosensors (ANNE™ Arc and ANNE™ Limb) with Bluetooth® 5 enabled and encrypted data communication to an iPad application. Study sensors to be applied on patients are:
  Sensor 1 - ANNE™ Arc with a Lithium-Polymer battery that contains a 6-axial inertial measurement unit (IMU), which includes a 3-axis gyroscope and 3-axis accelerometer, a power management component, an analog front-end component, passive electrodes for ECG, and bio-impedance feature that capture the following waveforms: heart rate (HR), respiratory rate (RR) and skin temperature.
  Sensor 2 - A limb unit (ANNE™ Limb) with embedded battery that captures the photoplethysmography (PPG) and SpO2 signals.
  Groups: Phase 1b
Device: ANNE™ Monitoring System (2 sensors) - version C — ANNE™ is a wireless vital sign monitoring device that uses soft, flexible, skin-mountable biosensors (ANNE™ Arc and ANNE™ Limb) with Bluetooth® 5 enabled and encrypted data communication to an iPad application. Study sensors to be applied on patients are:
  Sensor 1 - ANNE™ Arc with a Lithium-Polymer battery that contains a 6-axial inertial measurement unit (IMU), which includes a 3-axis gyroscope and 3-axis accelerometer, a power management component, an analog front-end component, passive electrodes for ECG, and bio-impedance feature that capture the following waveforms: heart rate (HR), respiratory rate (RR) and skin temperature.
  Sensor 2 - A limb unit (ANNE™ Limb) with embedded battery that captures the photoplethysmography (PPG) and SpO2 signals.
  Groups: Phase 2

SUMMARY:
The study will be conducted in a convenience sample of 75 infants admitted to the NICU at the Montreal Children's Hospital, divided into 3 phases: (a) Phase 1a - monitoring for 8h per day for 4 consecutive days, (b) Phase 1b - monitoring between 2h to 8h per day for 2 to 4 consecutive days, and (c) Phase 2- monitoring for 96h continuously.

Study objectives include:

1. Demonstrate the feasibility of continuous wireless monitoring in term and preterm infants with variable degrees of maturation and acuity in the NICU.
2. Assess safety of using a special wireless sensor system in neonates.
3. Evaluate the accuracy of proposed wireless technology as compared to standard monitoring technology in the NICU.

DETAILED DESCRIPTION:
Infants admitted in the NICU are all subject to continuous monitoring of vital signs such as heart rate, respirations and oxygen saturation (SpO2) by placing sensors, leads, or bands directly on infant's skin and connecting them to monitors via wires. However, despite the rapid technological advances in wireless monitoring and wearable devices across various industries, the health care sector has traditionally lagged. Therefore, the investigators aim to explore the safety and effectiveness of wireless monitoring (ANNE™ Monitoring System) and compare it with the traditional wired monitoring system on infants with variable degrees of maturity in the NICU.

More specifically, the investigators aim to examine (1) if it is feasible and to implement a wireless monitoring system in both term and preterm infants in the NICU; (2) if it is safe to use this particular wireless monitoring system among neonates; and (3) the accuracy of the wireless monitoring technology compared to the stand-of-care monitoring in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants in room air at enrollment
* Term infants with perinatal asphyxia undergoing therapeutic hypothermia at enrollment
* Healthy preterm infants in room air at enrollment
* Preterm infants on continuous positive airway pressure at enrollment
* Preterm infants on conventional mechanical ventilation at enrollment
* Preterm infants on high frequency ventilation at enrollment
* Preterm infants on nasal intermittent positive end expiratory pressure at enrollment
* Preterm infants on continuous positive airway pressure at enrollment

Exclusion Criteria:

* Congenital anomalies and surgical conditions (ex: gastroschisis, omphalocele, congenital diaphragmatic hernia)
* Congenital heart disorders
* Congenital skin infections or known conditions with fragile skin (such as epidermolysis bullosa)

Ages: 6 Hours to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants admitted to the NICU at the Montreal Children's Hospital with different levels of maturity/clinical conditions.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of wireless wearable heart rate data | 4 consecutive days of wireless monitoring
  Accuracy of wireless wearable heart rate data compared against the current standards of NICU bedside monitoring.
Accuracy of wireless wearable respiratory rate data | 4 consecutive days of wireless monitoring
  Accuracy of wireless wearable respiratory rate data compared against the current standards of NICU bedside monitoring.
Accuracy of wireless wearable skin temperature data | 4 consecutive days of wireless monitoring
  Accuracy of wireless wearable skin temperature data compared against the current standards of NICU bedside monitoring.
Accuracy of wireless wearable oxygen saturation (SpO2) data | 4 consecutive days of wireless monitoring
  Accuracy of wireless wearable SpO2 data compared against the current standards of NICU bedside monitoring.
Proportion of time exhibiting unreliable wireless device signals due to significant movement artifacts | 4 consecutive days of wireless monitoring
  Proportion of monitoring time exhibiting unreliable wireless device signals due to significant movement artifacts. The exact definition of unreliable for each of the signals will be outlined before study initiation.
Proportion of time with loss of network connections or other technical problems | 4 consecutive days of wireless monitoring
  Proportion of time with loss of network connections or other technical problems from the wireless wearables vs. the NICU bedside monitoring.
Skin integrity at the sites of sensor placement | 4 consecutive days of wireless monitoring
  Skin integrity at the site of wireless lead placements from de-identified digital photographs, evaluated by a board-certified dermatologist who will evaluate for signs of irritation, redness and/or erosions.
Evaluation of potential subjective pain experienced by infant at time of sensor removal | 4 consecutive days of wireless monitoring
  Assessing infants for presence of acute pain associated with sensor removal by administering Neonatal Infant Pain Scale (NIPS) at time of device removal.
Clinicians', nursing, and parental perceptions | 4 consecutive days of wireless monitoring
  Clinicians', nursing, and parental perceptions of the implementation of wireless wearable devices in the NICU.

SECONDARY OUTCOMES:
Automated reports of physiological health - electrocardiogram | 4 consecutive days of wireless monitoring
  Automated reports for electrocardiogram acquired from the wireless monitoring device
Automated reports of physiological health - respiratory waveforms | 4 consecutive days of wireless monitoring
  Automated reports for respiratory waveforms acquired from the wireless monitoring device
Automated reports of physiological health - oxygen saturation | 4 consecutive days of wireless monitoring
  Automated reports for oxygen saturation acquired from the wireless monitoring device
Automated reports of physiological health - temperature | 4 consecutive days of wireless monitoring
  Automated reports for temperature acquired from the wireless monitoring device
Comparison between chest and respiratory inductance plethysmography (RIP) and the wireless monitoring device | 2 to 3 consecutive hours each day during the 4-day continuous monitoring
  For patients in Cohort 2, we will compare the chest and abdominal wall movement signals derived from accelerometry with RIP (the gold standard) with the simultaneously recorded wireless monitoring device data.
Enhanced respiratory monitoring using accelerometry | 2 to 3 consecutive hours each day during the 4-day continuous monitoring
  For patients in Cohort 2, we will compare the chest and abdominal wall movement signals derived from accelerometry with thoracic impedance (the current standard) with the simultaneously recorded wireless monitoring device data.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Sant'Anna, MD PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Wissam Shalish, MD PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Robert E Kearney, PhD, Principal Investigator — McGill University
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada